CLINICAL TRIAL: NCT06266754
Title: The Non-Specific Immunological Effects of Providing Oral Polio Vaccine to Seniors in Guinea-Bissau
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OPV-IMMUNO-ADULT
Record Dates: First submitted 2024-01-18; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Vaccine Reaction
Keywords: Oral polio vaccine; Trained immunity
MeSH Terms: interventions — Poliovirus Vaccine, Oral

STUDY DESIGN:
Intervention Model Description: Randomised trial
Who Masked: Participant, Outcomes Assessor
Masking Description: A placebo will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral polio vaccine (Experimental): Oral polio vaccine, 2 drops on a sugar lump
  Interventions: Biological: Oral polio vaccine
- Placebo (Placebo Comparator): Saline, 2 drops on a sugar lump
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Oral polio vaccine — Standard oral polio vaccine
  Arms: Oral polio vaccine
Other: Placebo — Saline 0.9%
  Arms: Placebo

SUMMARY:
OPV is the live attenuated vaccine against polio virus. OPV has been key in almost eradicating polio infection. Intriguingly, OPV has been associated with lower all-cause mortality and morbidity. These beneficial OPV effects were seen in contexts with no circulating polio virus and thus have nothing to do with the specific effects of OPV against polio infection. They have been coined "non-specific effects" (NSEs). Such NSEs have also been observed for other live attenuated vaccines such as BCG vaccine and measles vaccine. The underlying immunological mechanisms are unknown. Other live vaccines with beneficial NSEs have been shown to induce epigenetic changes leading to "trained immunity". They have also been associated with decreased inflammation. In the present study it will be investigates whether OPV can induce trained immunity, reduce inflammation, and induce epigenetic modifications of the innate immune cells in senior citizens in Guinea-Bissau.

DETAILED DESCRIPTION:
The aim is to study the non-specific immunological effects of providing a single dose of OPV to seniors aged 50 and above in Guinea-Bissau:

Hypotheses

1. OPV induces innate immune training (substudy A)
2. OPV is associated with reduced systemic inflammation (substudy A)
3. OPV induces epigenetic modifications of the innate immune cells (substudy B)

Setting: Bandim Health Project (BHP)'s Health and Demographic Surveillance System (HDSS) in Bissau.

Design: Individually randomized trial in BHP's study area. Participants will be randomized 1:1 to OPV or placebo. To limit the amount of blood drawn from one single participant, two substudies with similar design will be conducted, with two different outcomes.

The outcomes of the two substudies will be as follows:

Substudy A: Immunological impact of OPV. Study the stimulation of cytokine production by heterologous stimuli as a biomarker of trained immunity induction and circulating biomarkers as a mirror of systemic inflammation induced by OPV.

Substudy B: Transcriptional and epigenetic reprogramming of immune cells by OPV. Study the transcriptional and epigenetic rewiring of immune cells induced by OPV by single-cell ATAC-Sequencing and RNA-Sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Living in a household which had a Bandim Health Project census visit conducted after 1 January 2017.
* Age above 50.
* Has a visible BCG scar.

Exclusion Criteria:

* Previous adverse events to OPV
* Suspicion of active viral/bacterial/HIV infection.

Ages: 50 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Levels of in vitro proinflammatory cytokines such as IL1-beta, TNF-alfa and IFN-gamma after stimulation of peripheral blood mononuclear cells with non-OPV antigens and mitogens | 1 month after the intervention
  Study the ability of cells of producing cytokines in vitro after heterologous stimuli. This is a well-established biomarker of trained immunity (ref: https://pubmed.ncbi.nlm.nih.gov/38198850/).
Levels of plasma markers of systemic inflammation such as TNF ligand superfamily member 12 (TWEAK) and sirtuin 2 (SIRT2) | 1 month after the intervention
  Study the effect on systemic inflammation induced by OPV. Previous studies have shown that BCG reduce up to a third of proinflammatory proteins as a marker of non-specific effects of that vaccine, we will study if this is the case also for OPV (ref:https://pubmed.ncbi.nlm.nih.gov/32692728/).
Amount of pseudo-bulk ATACseq and RNAseq - indicating chromatin accessibility of interferon-stimulated genes associated with the interferon response pathway in PBMCs. | 1 month after the intervention
  Study the epigenetic rewiring of immune cells induced by OPV by single-cell ATAC-Sequencing and whole-genome methylation assays. This is a new method to assess if there has been changes to the accessibility of the genes (ref: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9022455/).
Proportions of immune cell subsets | 1 month after the intervention
  Study the transcriptional effects of OPV on immune cell by studying the transcriptional rewiring of immune cells induced by OPV by single-cell RNA-Sequencing (ref: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9022455/).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie R Madsen, MD, PhD, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No
We collect sensitive data that cannot immediately be shared.